CLINICAL TRIAL: NCT05726058
Title: Ocular Blood Flow Imaging for Glaucoma Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Eye Institute (NEI) (NIH); Vasoptic Medical, Inc (Unknown)
Responsible Party: Principal Investigator, Osamah Saeedi, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00102645; 1R44EY034064-01 (NIH)
Record Dates: First submitted 2022-12-12; First posted 2023-02-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma
Keywords: glaucoma; xycam; blood flow; imaging; ophthalmology; retinal blood flow; eye disease
MeSH Terms: conditions — Glaucoma; Eye Diseases | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control (Other): All control participants will be first be imaged pre-intervention.
  Interventions: Device: XyCAM with oxygen
- Glaucoma (Other): All participants with glaucoma will be first be imaged pre-intervention.
  Interventions: Device: XyCAM with oxygen
- Pre-perimetric Glaucoma (Other): All participants with pre-perimetric glaucoma will be first be imaged pre-intervention.
  Interventions: Device: XyCAM with oxygen

INTERVENTIONS:
Device: XyCAM with oxygen — After the standard imaging protocols, participants will be asked to inhale 100% oxygen through a mask and will be re-imaged using the XyCAM RI or XyCAM FC.

SUMMARY:
The goal of this clinical trial is to investigate the use of an FDA-cleared retinal blood flow imaging instrument called the XyCAM RI and XyCAM FC (Vasoptic Medical, Inc., Columbia, MD) in glaucoma management.

The main question it aims to answer are:

* Can the investigators use blood flow to discriminate between eyes with early-stage glaucoma and variable-matched controls?
* Can the investigators validate that the XyCAM FC simultaneously captures both stereo fundus photography and ocular blood flow monitoring?

Participants will be

* measured for their blood pressure, heart rate, height, and weight
* dilated with tropicamide
* imaged using the XyCAM RI, fundus photography, optical coherence tomography, and standard automated perimetry
* imaged using the XyCAM RI while inhaling 100% oxygen through a mask

DETAILED DESCRIPTION:
The investigators will capture images of the participant's retina using the XyCAM RI or XyCAM FC ("test data") and by color fundus photography, optical coherence tomography (OCT), and standard automated perimetry (SAP) - the "standard clinical data". The investigators will perform five tests. The first two tests will be conducted using the XyCAM RI or XyCAM FC to obtain "test data". The final two tests will be conducted using routine clinical instruments to obtain "standard clinical data". The investigators will administer eye drops (Tropicamide) to dilate the participant's pupils prior to the first test. Tropicamide is a chemical that causes pupil dilation and is commonly used by doctors to examine the participant's eyes. The entire set of test data sessions should last less than eighty (80) minutes with an additional 60 minutes for carrying out the necessary procedures and imaging using the standard clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older with binocular vision
* Able to provide informed consent
* Patient is a healthy control OR is recommended for glaucoma assessment OR diagnosed with moderate to severe glaucoma in at least one eye as determined by Hodapp Anderson Criteria

Exclusion Criteria:

* The subject has significant media opacity (e.g., a visually significant cataract or significant corneal scar)
* The subject has previous ocular surgery other than uncomplicated cataract extraction, laser trabeculoplasty (ALT or SLT), or YAG capsulotomy
* The subject has prior ocular disease other than glaucoma
* The subject has anatomically narrow angles or a prior adverse reaction to administration of Tropicamide or fluorescein dye
* The subject has more than 15 diopters of refractive error
* The subject is a female who is pregnant or nursing
* The subject has diabetes mellitus

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Blood flow velocity measure | through study completion, an average of 1 year
  Dynamic video of ocular blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Grace Forbes, MS, Study Director — University of Maryland, Baltimore
Locations (1):
- University of Maryland Eye Associates at Redwood, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinnett A, Kandukuri J, Le C, Cho KA, Sinha A, Asanad S, Thompson G, Chen V, Rege A, Saeedi OJ. Dynamic Alterations in Blood Flow in Glaucoma Measured with Laser Speckle Contrast Imaging. Ophthalmol Glaucoma. 2022 May-Jun;5(3):250-261. doi: 10.1016/j.ogla.2021.10.005. Epub 2021 Oct 18. PMID 34673279